CLINICAL TRIAL: NCT02241005
Title: A Randomized Controlled Trial of the Safety and Efficacy of Theraworx Bath Wipes in the Reduction of Skin Colonization With Vancomycin-Resistant Enterococci Compared to Standard Bath Wipes in Children Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Theraworx Bath Wipes Versus Standard Bath Wipes in the Reduction of Vancomycin-Resistant Enterococci
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Avadim Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TWIPES; NCI-2015-00114 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Hematopoietic Stem Cell Transplantation; Vancomycin-Resistant Enterococci
Keywords: Health-care associated infection; Skin integrity; Antimicrobial resistance
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theraworx™ (Active Comparator): Participants are randomized to use the Theraworx™ bath wipes.
  Interventions: Other: Theraworx™ bath wipes
- Standard (Active Comparator): Participants are randomized to use standard bath wipes.
  Interventions: Other: Standard bath wipes

INTERVENTIONS:
Other: Theraworx™ bath wipes — Theraworx™ bath wipes will be supplied in packaging similar to the standard bath wipes used in this study. The bath wipes will be started on the day of admission, and used once daily for a period of 60 days post-HSCT.
  Arms: Theraworx™
Other: Standard bath wipes — Standard bath wipes will be supplied in packaging similar to the Theraworx™ bath wipes used in this study. The bath wipes will be started on the day of admission, and used once daily for a period of 60 days post-HSCT.
  Arms: Standard

SUMMARY:
Healthcare-associated infections (HAI) are associated with substantial morbidity, mortality and health-care costs in children undergoing hematopoietic stem cell transplantation (HSCT). These infections are often caused by a patient's own microbial flora. Hence reduction of microbes in the skin could lessen the risk of contamination of central venous catheters, Central Line Associated Blood-Stream Infections (CLABSI), and bacteremia due to compromise of skin integrity.

Theraworx™ (herein referred to as experimental wipes) is a self-drying, leave on cleansing agent that combines a specialized surfactant with skin healthy ingredients, including aloe, allantoin, vitamin E, and silver, which is the main antimicrobial ingredient. It can be used on all parts of the body including burns, abraded skin, and on patients with skin graft-versus-host-disease (GVHD). It is user friendly and obviates the risk of antimicrobial resistance. Microbiologic studies have shown several log fold reduction of bacteria including vancomycin-resistant enterococci, carbapenem resistant Escherichia coli, and activity against Staphylococcus aureus, Enterococcus faecalis, Clostridium difficile, Candida albicans, and viruses including influenza A and Herpes Simplex. There is no data regarding the use of Theraworx™ (experimental) bath wipes in children or the HSCT population.

Researchers at St. Jude Children's Research Hospital want to learn if daily bathing with experimental bath wipes will be well tolerated and associated with reduction in microbial skin colonization in this population.

DETAILED DESCRIPTION:
Participants will be randomized to receive either a daily bath with the experimental bath wipes, or the standard bath wipes, beginning on the day of admission, and to be used once daily for a period of 60 days post-HSCT. In the first 12 patients randomized to the experimental wipes, if no patient has grade IV skin toxicity that is attributable to the experimental wipes, then the trial will continue until a total of 250 evaluable participants have been enrolled. Assessment of skin colonization will be performed before admission, at the time of discharge, and post-HSCT.

Randomization will take place at the time the participant is enrolled and will be performed by staff within the Nursing Research Department. Participants will be assigned to either experimental or standard bath wipes in a 1:1 ratio. Randomization may be stratified for nature of transplant (autologous vs. allogeneic); and in the case of allogeneic transplant stratified for total body irradiation vs. no total body irradiation. The investigators, practicing clinician and the clinical research staff will remain blinded to the treatment.

PRIMARY OBJECTIVES:

* Assess the safety of the experimental bath wipes in 12 patients.
* Assess the skin colonization with vancomycin-resistant enterococci in patients using the experimental wipes compared to standard bath wipes.

SECONDARY OBJECTIVES:

* Assess skin colonization with bacterial pathogens.
* Compare the skin colonization with multi-drug resistant organisms (MRDO) and central line-associated bloodstream infection (CLABSI) rates.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 21 years of age.
* Scheduled to undergo either autologous or allogeneic hematopoietic stem cell transplant

Exclusion Criteria:

* Participant/Parent/Legally authorized representative (LAR) unwilling to give written informed consent.
* (Female only) Known pregnancy (negative serum or urine pregnancy test to be conducted within 14 days prior to enrollment).
* (Female only) Breast feeding

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2014-10-30 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients using Theraworx™ wipes who experience any grade IV skin toxicity | Through date of discharge from inpatient unit, or maximum of 60 days after study enrollment
  In the first 12 evaluable patients in the Theraworx™ arm of the randomized controlled trial, we will closely monitor for the safety of experimental bath wipes. Since no grade IV toxicity attributable to the wipes is expected in the standard bath wipes arm, if at any time during the study in the first 12 evaluable participants in the experimental arm we observe one patient with grade IV skin rash toxicity in the experimental arm which is attributable to the experimental bath wipes , then the study will be stopped and the use of experimental bath wipes for HSCT patients will be considered unsafe. If the use of experimental bath wipes for HSCT patients is considered feasible, the trial will continue. 95% Blyth-Still-Casella will be provided.
Proportion of patients with vancomycin-resistant enterococci (VRE) colonization by study arm | At enrollment, at the time of initial discharge from the inpatient unit, and at end of study (60 days)
  The proportion of patients with VRE colonization at enrollment and at the time of initial discharge from the inpatient unit in the groups of patients using the experimental and standard bath wipes and their 95% confidence intervals (CI) will be provided. Fisher's exact test will be used to test for the null hypothesis that two proportions are equal

SECONDARY OUTCOMES:
Number of different bacterial species in participants by study arm | At enrollment, at the time of initial discharge from the inpatient unit, and at end of study (60 days)
  Summary statistics for the number of different bacterial species in groups of patients using the experimental and standard bath wipes will be provided. Exact Wilcoxon rank sum test will be used to compare the medians of the numbers of different bacterial species in two groups.
Proportion of patients with multi-drug resistant organisms (MRDO) and central line-associated bloodstream infection (CLABSI) | At enrollment, at the time of initial discharge from the inpatient unit, and at end of study (60 days)
  The proportions of patients with MRDO and CLABSI in the groups of patients using the experimental wipes and standard bath wipes and their 95% Blyth-Still-Casella (BSC) CIs will be provided. Fisher's exact test will be used to test for the null hypothesis that two proportions are equal.

CONTACTS AND LOCATIONS:
Overall Officials: Margie Kjellin, RN, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols